CLINICAL TRIAL: NCT03250455
Title: Prognostic Value of CT dynamIc Myocardial Perfusion in Patients With Obstructive Coronary Artery Stenosis
Acronym: VALIDITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Guangdong Provincial People's Hospital (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Bin Lu, chief of Radilogy, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CIFuwaiHospital-2
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: CT Perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CTA+CTP
  Interventions: Diagnostic Test: CTA CTP
- CTA only
  Interventions: Diagnostic Test: CTA

INTERVENTIONS:
Diagnostic Test: CTA CTP — CT Angiography myocardial CT Perfusion
  Groups: CTA+CTP
Diagnostic Test: CTA — CT Angiography
  Groups: CTA only

SUMMARY:
VALIDITY is a prospective, open-label, multicenter, randomized controlled trial （ClinicalTrials.gov number）. The study was designed to evaluate the value of noninvasive anatomic CTA combined with functional CTP for the next clinical decision making and the added prognostic value of CTP beyond CTA.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years.
2. stable chest pain with obstructive coronary stenosis (50-90%) assessed by CTA.

Exclusion Criteria:

* (1) Diagnosed or suspected acute coronary syndrome (ACS) requiring hospitalization or urgent or emergent testing; Elevated troponin or creatine kinase-myocardial band (CK-MB).

  (2) Hemodynamically or clinically unstable condition systolic blood pressure (BP) < 90 mmHg, atrial or ventricular arrhythmias, or persistent resting chest pain felt to be ischemic despite adequate therapy.

  (3) Known CAD with prior Myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG).

  (4) Known significant congenital, valvular (> moderate) or cardiomyopathic process (hypertrophic cardiomyopathy or reduced systolic left ventricular function (LVEF) ≤ 40%)) which could explain cardiac symptoms.

  (5) Contraindication to undergoing CTA, including but not limited to: a. Allergy to iodinated contrast agent, b. Unable to receive beta blockers, c. creatinine ≥1.7 mg/dl or GFR≤30 ml/min , d. Pregnancy.

  (6) Contraindication to ATP, including but not limited to: a. II or III atrioventricular block, b. bronchial asthma, c. hypotension (SBP<90mmHg), d. bronchial stenosis or bronchospasm, e. acute myocardial infarction, f. left main stenosis, g. unstable angina, h. allergy to aminophylline.

  (7) Life expectancy < 2 years. (8) Unable to provide written informed consent or participate in long-term follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stable chest pain and diagnosed of obstructive coronary stenosis (50-90%) by CTA were enrolled.
Sampling Method: Probability Sample
Enrollment: 1748 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 90 days, 6 months, 12 months, 24 months and 36 months
  death, myocardial infarction and unstable angina requiring hospitalization

SECONDARY OUTCOMES:
invasive coronary angiography and revascularization | 90 days, 6 months, 12 months, 24 months and 36 months
  invasive coronary angiography and PCI or CABG
he incidence of a composite of major complications from cardiovascular procedures and testing | 90 days, 6 months, 12 months, 24 months and 36 months
  stroke, bleeding, anaphylaxis, renal failure
Quality of Life | 90 days, 6 months, 12 months, 24 months and 36
  Quality of Life (QOL) as Measured by Seattle Angina Scale Anginal Frequency Subscale
total medical cost | 90 days and 3 years
  Assess and compare total medical cost for the two diagnostic testing arms by intention to treat

CONTACTS AND LOCATIONS:
Overall Officials: Bin Lu, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (5):
- China (5):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Xiehe Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Shanghai Sixth People's Hospital, Shanghai
  - General hospital of tianjin medical university, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided